CLINICAL TRIAL: NCT06097286
Title: A Comparative Study Between Ultrasound Guided External Oblique Intercostal Plane (EOIP) Block and Erector Spinae Plane (ESP) Block for Postoperative Analgesia in Upper Abdominal Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MD80/2023
Record Dates: First submitted 2023-09-21; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-03

CONDITIONS: Block
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- external oblique intercostal plane block (Active Comparator)
  Interventions: Procedure: external oblique intercostal plane block
- erector spinae plane block (Active Comparator)
  Interventions: Procedure: erector spinae plane block
- control group (No Intervention)

INTERVENTIONS:
Procedure: external oblique intercostal plane block — o EOIP Group (ŋ=25): Patients will receive ultrasound guided External oblique intercostal plane block with 20 ml of LA mixture (10 mL of bupivacaine 0.5%, 5 mL of lidocaine 2% and 5 mL of normal saline to make a total volume of 20 ml.) at the end of procedure, unilaterally or bilaterally according to the surgery.
  Arms: external oblique intercostal plane block
Procedure: erector spinae plane block — o ESP Group (ŋ=25): Patients will receive ultrasound guided Erector spinae plane block with 20 ml of LA mixture (10 mL of bupivacaine 0.5%, 5 mL of lidocaine 2% and 5 mL of normal saline to make a total volume of 20 ml.) at the end of procedure, unilaterally or bilaterally according to the surgery.
  Arms: erector spinae plane block

SUMMARY:
Upper abdominal incisions, such as the oblique subcostal laparotomy, can cause severe pain and can lead to significant respiratory impairment.

Erector spinae plane (ESP) block is the deposition of local anaesthetic (LA) in the interfascial plane at the paraspinal region. It provides effective visceral and somatic analgesia.

External oblique intercostal plane (EOIP) block is a newly described block at which local anaesthetic (LA) is deposited in the interfascial plane deep to external oblique muscle at the sixth intercostal space. It provides blockade of the thoracoabdominal nerves at the level of T6 to T10.

In this study, the investigators compare between ultrasound (US) guided external oblique intercostal plane block and erector spinae plane block, in providing postoperative analgesia for upper abdominal surgeries

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Society of Anesthesiologists physical status (ASA) I and II.
* Both sex.
* 20 to 60 years old patients.
* upper abdominal surgeries.

Exclusion Criteria:

* Refusal of the patient to consent.
* Patients with ASA status III or IV
* Patients with bleeding disorders and coagulopathy (INR≥1.6 & PTT≥50 sec).
* Infection at the injection site.
* Allergy to local anesthetics.
* Patients with ages less than 20 or more than 60
* Patients with pre-existing myopathy or neuropathy.
* Patients with chronic pain syndromes.
* Patients with history of long acting opioids or steroids preoperatively.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
amount of total 24 hour pethidine consumption (mg) . | 24 hours postoperatively
  to measure total 24 hour pethidine consumption postoperatively.

SECONDARY OUTCOMES:
visual analogue scale (VAS) at rest and movement. | 24 hours postoperatively
  recorded postoperative immediately and 2, 4, 6, 8, 12, 18 and 24 hours. The Visual Analogue Scale (VAS) measures pain intensity. The visual analogue scale (VAS) consists of a 10 cm line, with two end points representing 0 (no pain) and 10 (pain as bad as it could possibly be).
mean arterial blood pressure (MAP) | 24 hours postoperatively
  recorded postoperative immediately and 2, 4, 6, 8, 12, 18 and 24 hours
heart rate (HR) | 24 hours postoperatively
  recorded postoperative immediately and 2, 4, 6, 8, 12, 18 and 24 hours
incidence of postoperative complications (nausea and vomiting) | 24 hours postoperatively
  recorded postoperative immediately and 2, 4, 6, 8, 12, 18 and 24 hours
time to start mobilization | 24 hours postoperatively
  recorded postoperative immediately and 2, 4, 6, 8, 12, 18 and 24 hours